CLINICAL TRIAL: NCT00981981
Title: Effect of Varying Dose and Molecular Weight on the Serum LDL-cholesterol-lowering Properties of Oat β-glucan
Brief Title: Effect of the Molecular Weight of Oat β-glucan on Its Ability to Lower Serum Cholesterol
Acronym: Bluebird
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glycemic Index Laboratories, Inc (Industry)
Collaborators: CreaNutrition, AG (Unknown); University of Guelph (Other); University of Sydney (Other); Laval University (Other); Reading Scientific Services Ltd. (Industry); University of Toronto (Other); Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Thomas MS Wolever, President, Glycemic Index Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIL8034
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Hypercholesterolemia
Keywords: humans; randomized clinical trial; dietary fiber; nutrition; beta-glucan; oats; LDL cholesterol; coronary heart disease
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control (Placebo Comparator): Wheat bran cereal
  Interventions: Dietary Supplement: Wheat bran
- 3g high MW (Active Comparator): Cereal containing 3g high molecular weight oat beta glucan
  Interventions: Dietary Supplement: 3g high MW
- 4g medium MW (Active Comparator): Cereal containing 4g oat beta glucan with medium molecular weight
  Interventions: Dietary Supplement: 4g medium MW
- 3g medium MW (Active Comparator): Cereal containing 3g oat beta glucan with medium molecular weight
  Interventions: Dietary Supplement: 3g medium MW
- 4g low MW (Active Comparator): Cereal containing 4g oat beta glucan with low molecular weight
  Interventions: Dietary Supplement: 4g low MW

INTERVENTIONS:
Dietary Supplement: Wheat bran — 21g per day of ready to eat breakfast cereal containing wheat bran with 8g of total dietary fiber and 0.5g beta-glucan.
  Arms: Control
Dietary Supplement: 3g high MW — 20.2 grams per day of ready to eat cereal containing 6g total dietary fiber and 3g oat beta glucan with high molecular weight
  Arms: 3g high MW
Dietary Supplement: 4g medium MW — 28.5g ready to eat cereal containing 8g total dietary fiber and 4g oat beta glucan with medium molecular weight
  Arms: 4g medium MW
Dietary Supplement: 3g medium MW — 21.1g of ready to eat cereal containing 6g total fiber and 3g oat beta glucan with a medium molecular weight
  Arms: 3g medium MW
Dietary Supplement: 4g low MW — 28.7g ready to eat cereal containing 8g total dietary fiber and 4g oat beta glucan with low molecular weight
  Arms: 4g low MW

SUMMARY:
The purposes of this study were:

1. To determine if a breakfast cereal containing 3g of high molecular weight oat beta-glucan fiber would lower low-density lipoprotein (LDL) - cholesterol (the "bad" cholesterol) compared to a control cereal containing wheat fiber.
2. To determine if the LDL-cholesterol-lowering effect of oat beta-glucan fiber was reduced when the molecular weight of the fiber was reduced.

DETAILED DESCRIPTION:
The FDA allows a health claim that oat products may reduce the risk of heart disease, based on meta-analyses showing a cholesterol-lowering effect of oat beta-glucan, if the product delivers at least a 3g daily dose of oat beta-glucan. However, not all studies have demonstrated a lowering of oat products. This may be due to variable bioactivity of the beta-glucan in the oat products. The bioactivity of oat beta-glucan is believed to depend upon its viscosity in the gut. Factors influencing viscosity include the molecular weight (MW) of the beta-glucan molecule and the amount of soluble beta-glucan in the product, which, in turn determines its concentration (C) in solution. In finished food products both MW and C can be modified by beta-glucanase enzymes present in other ingredients in the food (eg. wheat flour), processing (eg. extrusion) and storage (eg. freezing of moist products such as muffins). The effect of altering the MW and solubility of beta-glucan in foods on glycemic responses has been shown, but a role for MW and C in cholesterol lowering has not been established.

To address this issue, this study was designed with 2 primary objectives:

1. An extruded oat cereal containing 3g high-molecular weight oat β-glucan daily will reduce LDL cholesterol compared to a control wheat bran cereal.
2. A significant correlation exists between LDL cholesterol and log(C×MW), where C is the amount of soluble β-glucan in the daily dose of cereal and MW is the molecular weight of the β-glucan in the cereal.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 18.5 to 40.0 kg/m^2
* no intention to lose or gain weight
* fasting total cholesterol 5.0 to 8.0 mmol/L
* fasting LDL cholesterol 3.0 to 5.0 mmol/L
* consuming diet containing <15% energy from saturated fat

Exclusion Criteria:

* use of any cholesterol-lowering drug, herbal or nutritional supplement
* regular consumption of oatmeal, oat bran or psyllium - containing cereals
* fasting serum triglycerides >4.0mmol/L
* serum aspartate transaminase >1.5 times upper limit of normal
* serum urea or creatinine >1.8 times upper limit of normal
* presence of diabetes or fasting glucose >6.9mmol/L
* presence or recent major surgical or medical event
* allergy to wheat or oats
* presence of condition or drug which alters digestion or absorption of foods

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Serum LDL-cholesterol lowering effect of 3g high MW beta-glucan | 4 weeks
Correlation between serum LDL-cholesterol lowering and log(MW*C) | 4 weeks

SECONDARY OUTCOMES:
Total cholesterol | 4 weeks
Serum triglycerides | 4 weeks
Serum HDL cholesterol | 4 weeks
Fasting serum glucose | 4 weeks
Serum aspartate transaminase | 4 weeks
serum c-reactive protein | 4 weeks
Serum urea | 4 weeks
Serum creatinine | 4 weeks
Time course of changes in blood lipids | 4 weeks
Blood pressure | 4 weeks
Macronutrient composition of diet | 4 weeks
Symptoms questionnaire | 4 weeks
apolipoprotein B | 4 weeks
Serum markers of cholesterol absorption and synthesis | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — Glycemic Index Laboratories, Inc; Peter J Wood, PhD, Study Director — Agriculture and Agri-Food Canada; Susan M Tosh, PhD, Study Director — Agriculture and Agri-Food Canada; Alison L Gibbs, PhD, Study Director — Department of Statistics, University of Toronto
Locations (5):
- SUGiRS Human Nutrition Unit, School of Molecular & Microbial Biosciences, Unviersity of Sydney, Sydney, New South Wales, Australia
- Canada (3):
  - Human Nutraceutical Research Unit, Department of Human Health and Nutritional Sciences, University of Guelph, Guelph, Ontario
  - Glycemic Index Laboratories, Inc., Toronto, Ontario
  - Nutraceuticals and Functional Foods Institute, Faculte des science de l'agriculture et de l'alimentation, Universite Laval, Laval, Quebec
- Reading Scientific Services, Ltd (RSSL), Reading, Berkshire, United Kingdom

REFERENCES:
- [Result] Wolever TM, Tosh SM, Gibbs AL, Brand-Miller J, Duncan AM, Hart V, Lamarche B, Thomson BA, Duss R, Wood PJ. Physicochemical properties of oat beta-glucan influence its ability to reduce serum LDL cholesterol in humans: a randomized clinical trial. Am J Clin Nutr. 2010 Oct;92(4):723-32. doi: 10.3945/ajcn.2010.29174. Epub 2010 Jul 21. PMID 20660224
- [Result] Tosh SM, Brummer Y, Miller SS, Regand A, Defelice C, Duss R, Wolever TM, Wood PJ. Processing affects the physicochemical properties of beta-glucan in oat bran cereal. J Agric Food Chem. 2010 Jul 14;58(13):7723-30. doi: 10.1021/jf904553u. PMID 20527967
- [Derived] Wolever TM, Gibbs AL, Brand-Miller J, Duncan AM, Hart V, Lamarche B, Tosh SM, Duss R. Bioactive oat beta-glucan reduces LDL cholesterol in Caucasians and non-Caucasians. Nutr J. 2011 Nov 25;10:130. doi: 10.1186/1475-2891-10-130. PMID 22118569